CLINICAL TRIAL: NCT02862041
Title: Role of Echogenic Versus Nonechogenic Needles in Ultrasound Guided Infraclavicular Brachial Plexus Block Success Rate: A Comparative Study
Brief Title: Effectiveness of Echogenic and Nonechogenic Needles in Ultrasound Guided Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Vinoth Kumar, Junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NK/1609/MD/10109-10
Record Dates: First submitted 2016-06-28; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Upper Extremity Injury Trauma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Echogenic (Active Comparator): Ultrasound guided infraclavicular brachial plexus block with Pajunk sonoplex echogenic needle
  Interventions: Device: Echogenic needle - Pajunk sonoplex echogenic needle
- Group Nonechogenic (Placebo Comparator): Non echogenic needle group, ultrasound guided infraclavicular brachial plexus block with Stimuplex Braun non echogenic needle
  Interventions: Device: Non Echogenic needle - Stimuplex Braun Nonechogenic needle

INTERVENTIONS:
Device: Echogenic needle - Pajunk sonoplex echogenic needle — Ultrasound guided infraclavicular brachial plexus block for upper extremity surgeries
  Arms: Group Echogenic
Device: Non Echogenic needle - Stimuplex Braun Nonechogenic needle — Ultrasound guided infraclavicular brachial plexus block for upper extremity surgeries
  Arms: Group Nonechogenic

SUMMARY:
In this prospective, randomized, double blinded study, the needle tip and needle shaft visibility of echogenic and nonechogenic needle were compared in ultrasound guided infraclavicular brachial plexus block. Sixty patients scheduled for upper extremity surgery were included in the study. Patients were randomised into two groups, group E (Echogenic) and group NE (Nonechogenic) with 30 subjects in each group. Under ultrasound guidance infraclavicular brachial plexus block was performed. In Group E, Pajunk Sonoplex echogenic needle was used and in Group NE, Stimuplex Braun nonechogenic needle was used. The subjective assessment for needle tip/shaft visibility as scored by the performer and the objective assessment from the recorded block procedure video were noted.

DETAILED DESCRIPTION:
The aim of the investigators study was to find out the better among the echogenic and nonechogenic needle in needle tip/shaft visibility and the block success rate in ultrasound guided infraclavicular brachial plexus block. Sixty patients were randomized into two groups, Group E (echogenic group) and Group NE (nonechogenic group) with thirty patients in each group. The ultrasound imaging of each nerve block was video recorded for later analysis. Recording commenced from skin puncture and stopped at the time of final needle removal (total block time). After each block the performer was asked to subjectively score the percentage time he had visualized the needle tip and needle shaft on a 5 point scale (1 = 0%-20%, 2 = 20%-40%, 3 = 40%- 60%, 4 = 60%-80%, 5 = 80%-100%). The recorded video was later analysed by an investigator. An objective measurement of percentage needle tip visibility and needle shaft visibility was calculated for each nerve block using the formula,

Time in view (needle tip) / total block time x 100

Time in view (needle shaft) / total block time x 100

The subjective assessment for needle tip/shaft visibility as scored by the performer and the objective assessment from the recorded block procedure video were noted. Other block parameters were also compared.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years, both male and female scheduled for upper extremity surgery

Exclusion Criteria:

* Clinically significant coagulopathy
* Local anesthetic allergy
* Preexisting motor or sensory deficit in the operative limb
* Uncontrolled hypertension and unstable Ischemic Heart disease
* Body mass index > 35
* Patients who needs general anaesthesia for surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Needle tip and shaft visibility | Duration of Block procedure
  Percentage Needle Tip & shaft visibility calculated using the formula - Time in view (needle tip or shaft) / total block time*100

SECONDARY OUTCOMES:
Duration of block procedure | 5- 15 minutes. Start of skin puncture till the final needle removal
Time to onset of sensory blockade | 0- 15minutes. Time (Minutes) between finishing injection of Local anaesthetic and to no response to pin prick test.
Time to onset of motor blockade | 0- 20 minutes. Time (Minutes) between finishing injection of Local anaesthetic and onset of full paralysis.
Duration of sensory blockade | 0- 6 hours. Time (Hours) between the block completion and the first pain postoperatively.
Duration of motor blockade | 0- 5 hours. Time (Hours) between the full paralysis and recovery of motor functions.
Block success rate of echogenic and Nonechogenic group. | Duration of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vinoth kumar, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hebard S, Hocking G. Echogenic technology can improve needle visibility during ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2011 Mar-Apr;36(2):185-9. doi: 10.1097/aap.0b013e31820d4349. PMID 21425515
- [Background] Duger C, Isbir AC, Kaygusuz K, Ozdemir Kol I, Gursoy S, Ozturk H, Mimaroglu C. The importance of needle echogenity in ultrasound guided axillary brachial plexus block: a randomized controlled clinical study. Int J Med Sci. 2013 Jul 4;10(9):1108-12. doi: 10.7150/ijms.6598. Print 2013. PMID 23869186